CLINICAL TRIAL: NCT01747681
Title: Results at 10 to 14 Years After Microfracture in Articular Cartilage Defects in the Knee
Brief Title: Results at 10 to 14 Years After Microfracture in the Knee
Status: Completed | Type: Observational
Sponsor: Bergen Orthopedic Study Group (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-Microfracture
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Articular Chondral Defect
Keywords: chondral defect; microfracture; arthroscopy; cartilage repair; outcome study; Lysholm score
MeSH Terms: conditions — Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Microfracture: Microfracture of articular chondral defect
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Procedure: Microfracture

SUMMARY:
Articular cartilage lesions are commonly occurring. In a prospective study of 1,000 knee arthroscopies focal chondral or osteochondral defects were found in 19% of the patients (Hjelle 2002). Chronic articular cartilage defects do not heal spontaneously. However, acute traumatic osteochondral lesions or surgically inflicted lesions extending into subchondral bone, e.g. by drilling (Pridie 1959), spongialization, abrasion or microfracture with an angled awl (Rodrigo 1994) causing the release of pluripotent mesenchymal stem cells from the bone marrow, may heal with repair tissue consisting of fibrous tissue, fibrocartilage or hyaline-like cartilage. The microfracture technique causes little damage to the subchondral bone plate and the risk of heat necroses caused by drilling or abrasion is eliminated. The quality of the repair tissue after these bone marrow stimulating techniques depends on various factors including the species and age of the individual, the size and localization of the defect, the surgical technique, e.g., how the subchondral bone plate is treated, and the postoperative rehabilitation protocol. Microfracture has been used in small traumatic defects in young sporting individuals (Steadman 2003) as well as in larger osteoarthritic lesions in older patients (Miller 2004, Steadman 2007). The purpose of the present study was to investigate the long-term clinical outcome 10 to 14 years after microfracture of articular cartilage defects in the knee and possible predictors of good and poor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic focal full-thickness chondral lesions verified by arthroscopic examination and a minimum of 10-year follow-up.

Exclusion Criteria:

* Exclusion criteria were joint space narrowing (< 4 mm) on standard antero-posterior x-ray films,
* axial malpositioning,
* ligament instabilities or inability to follow the rehabilitation protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients operated with a microfracture of articular chondral defects in the knee at the Deaconess University Hospital from 1999 to 2002.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Lysholm knee score | 10 to 14 years after surgery (in 2012-2013)
  All patients operated with a microfracture chondroplasty in the knee in 1999-2002 are invited to complete a patient-administered Lysholm score form

CONTACTS AND LOCATIONS:
Overall Officials: Eirik Eirik, MD, PhD, Study Director — Professor
Locations (1):
- Deaconess University Hospital, Haraldsplass, Bergen, Hordaland, Norway

REFERENCES:
- [Result] Solheim E, Hegna J, Inderhaug E, Oyen J, Harlem T, Strand T. Results at 10-14 years after microfracture treatment of articular cartilage defects in the knee. Knee Surg Sports Traumatol Arthrosc. 2016 May;24(5):1587-93. doi: 10.1007/s00167-014-3443-1. Epub 2014 Nov 23. PMID 25416965